CLINICAL TRIAL: NCT07343089
Title: A Multicenter Real-life Study of Disseminated Borreliosis Cases Occurring in Patients Receiving Anti-CD20 Treatment in France
Acronym: BorDiMab
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9819
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Borrelia Infections
Keywords: Borreliosis, Lyme; Borrelia Infections; Borrelia Burgdorferi; Borrelia Miyamotoi; Anti-CD20 monoclonal antibodies
MeSH Terms: conditions — Borrelia Infections; Lyme Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical, biological, radiological, and pharmacological description of cases of disseminated borreliosis (Borrelia burgdorferi sl. and Borrelia miyamotoi) occurring in patients who received drug treatment based on anti-CD20 monoclonal antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Minor or adult subject
* Having presented disseminated borreliosis confirmed by molecular biology (Borrelia burgdorferi sl. or Borrelia miyamotoi) within 24 months of receiving treatment with an anti-CD20 monoclonal antibody between January 1, 2010, and July 30, 2025.

Exclusion Criteria:

- Refusal to participate in the study

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient having presented disseminated borreliosis confirmed by molecular biology (Borrelia burgdorferi sl. or Borrelia miyamotoi) within 24 months of receiving treatment with an anti-CD20 monoclonal antibody between January 1, 2010, and July 30, 2025.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-29 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08-29 (Estimated)

PRIMARY OUTCOMES:
Description of the clinical presentation of cases of disseminated borreliosis occurring in patients receiving anti-CD20 therapy in France | Up to 12 months
  The clinical presentation describes how the disease manifests in patients:
  * the symptoms,
  * their severity,
  * and their progression.
  Example:
  Two patients may have the same disease, but one will primarily experience fever while the other will have neurological symptoms. This is part of the clinical presentation.

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratoire de Bactériologie - CHU de Strasbourg - France, Strasbourg, France